CLINICAL TRIAL: NCT05193994
Title: Randomised Double-Blind Placebo-Controlled Phase 3 Trial of Triumeq in Amyotrophic Lateral Sclerosis
Brief Title: Triumeq in Amyotrophic Lateral Sclerosis
Acronym: LIGHTHOUSE II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A planned interim analysis resulted in the recommendation that the trial be stopped. The results showed no benefit of Triumeq for people with ALS compared with placebo on survival, the primary outcome measure.
Sponsor: Macquarie University, Australia (Other)
Collaborators: King's College London (Other); Stichting TRICALS Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIGHTHOUSE II; 2020-005069-15 (EudraCT Number)
Record Dates: First submitted 2021-12-06; First posted 2022-01-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 2:1 ratio to receive either triumeq or placebo
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dolutegravir/Abacavir/Lamivudine (Experimental): Combination of Dolutegravir, Abacavir and Lamivudine in a single product/capsule.
  4 capsules to be taken orally once daily (all 4 at the same time, each capsule is Dolutegravir 12.5mg, Abacavir 150mg and Lamivudine 75mg). Maximum duration is 24months
  Interventions: Drug: Dolutegravir, Abacavir and Lamivudine
- Placebo (Placebo Comparator): 4 capsules to be taken orally once daily (all 4 at the same time). Maximum duration is 24months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dolutegravir, Abacavir and Lamivudine — Dolutegravir 50mg, Abacavir 600mg and Lamivudine 300mg.
  Other Names: Triumeq
  Arms: Dolutegravir/Abacavir/Lamivudine
Drug: Placebo — Matching placebo.
  Arms: Placebo

SUMMARY:
To determine if Triumeq improves survival in Amyotrophic Lateral Sclerosis (ALS) compared with placebo

DETAILED DESCRIPTION:
This Randomised Double-Blind Placebo Controlled trial seeks to investigate whether the combination medicine Triumeq (dolutegravir 50mg, abacavir 600mg, lamivudine 300mg), already sold in Australia for HIV treatment is effective in delaying progression of theAmyotrophic Lateral Sclerosis (ALS) disease and if it is safe and well tolerated in patients with ALS. This medication is very commonly prescribed for patients with HIV. The secondary aim of this study is to assess patient's health outcomes whilst taking this medication for their ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of screening
2. Diagnosis of ALS according to the Gold Coast Criteria
3. Capable of providing informed consent and complying with trial procedures
4. TRICALS risk profile > -6.0 and < -2.0
5. Those taking Riluzole must be on a stable dose for at least 30 days prior to the baseline visit or must have stopped taking Riluzole at least 30 days prior to the baseline visit
6. Women must not become pregnant (e.g., post-menopausal, surgically sterile, using highly effective birth control methods or not having potentially reproductive sex) for the duration of the study plus five days. Highly effective methods of birth control are those with a failure rate of < 1% per year when employed consistently and correctly, e.g. Combined (oestrogen and progestogen containing) hormonal contraception or progestogen-only hormonal contraception. For more information, please refer to the HMA CTFG Guidelines: https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf?fbclid=IwAR3AY5Ha0ESDyqIBeUaYI9VTFWmx9bbt8NZ-80N-5ME6pkBb1UHvFsTwqlQ
7. Women of childbearing potential must have a negative serum pregnancy test at screening and be non-lactating. Patients will be advised regarding appropriate contraception. A menstruation history will be taken at each visit. Women of childbearing potential are defined as females who are fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy (https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf?fbclid=IwAR3AY5Ha0ESDyqIBeUaYI9VTFWmx9bbt8NZ-80N-5ME6pkBb1UHvFsTwqlQ)
8. For participants taking antacids (regularly or as required), participant is willing and able to avoid taking antacids for at least 6 hours before and 2 hours after Triumeq
9. Participant taking taurursodiol supplements (TUDCA) can participate in this trial if the supplement does not contain sodium phenylbutyrate.
10. Participants taking taurursodiol supplements (TUDCA) that also contain sodium phenylbutyrate must be willing to stop supplementation 30 days prior randomisation.

Exclusion Criteria:

1. People who are HLA-B*5701 positive
2. Known hypersensitivity to Dolutegravir, Abacavir or Lamivudine, or to any of the excipients
3. Safety Laboratory Criteria at screening:

   * ALT ≥ 5 times upper limit of normal (ULN)
   * AST ≥ 3 times ULN
   * Bilirubin ≥ 1.5 times ULN with clinical indicators of liver disease
   * Creatinine clearance < 30 mL / min
   * Platelet concentration of < 100 x109 per L
   * Absolute neutrophil count of < 1x109 per L
   * Haemoglobin < 100 g/L
   * Amylase ≥ 2 times ULN
   * Lactate ≥ 2 times ULN
4. Moderate to severe hepatic impairment, as defined by local clinical guidelines
5. Presence of HIV antibodies at screening
6. Presence of Hepatitis C antibodies at screening unless participants have had effective treatment for Hepatitis C
7. Presence of Hepatitis B core or surface antigen at screening
8. Participation in any other investigational drug trial or using investigational drug within 30 days prior to screening
9. Use of NIV ≥22 h per day or having a tracheostomy
10. Edaravone dose within 30 days prior to screening. Edaravone is approved by the FDA and in Japan, but remains an investigational product in Europe and Australia
11. Clinically significant history of unstable or severe cardiac, oncological, psychiatric, hepatic, or renal disease or other medically significant illness
12. Taking medication contraindicated with Triumeq: Dofetilideor Fampridine (dalfampridine)
13. Taking Tofersen within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Measure overall survival at 24 months or after a minimum of 212 events | 24 months
  Overall survival is measured as death from any cause, in participants with ALS at 24 months, or after a minimum of 212 events.

SECONDARY OUTCOMES:
Measure scoring in the ALS-Functional Rating Scale Revised (ALSFRS-R) at 3 monthly intervals. | 24 months
  The ALSFRS-R is a 12 item participant self-report measure that monitors ALS disease progression, where a higher score reflects a better outcome.
Number of participants with abnormal Slow Vital Capacity measured by hand spirometry at 3 monthly intervals | 24 months
  Slow vital capacity is measured in litres, and as a % of predicted.
Measure plasma creatinine at 3 monthly intervals | 24 months
  Plasma creatinine is assessed to monitor kidney function
Assign a value using the King's Staging Scale to describe degree of disease advancement over time | 24 months
  The King's Staging Scale is a clinical staging system defining four stages of ALS assessed by way of a semi-structured interview with the participant.
Evaluate the incidence of treatment-emergent adverse events | 24 months
  based on physical examinations and patient reported symptoms.
Measure study medication discontinuation | 24 months
  the number of participants who discontinue study medication will be assessed to assess tolerability
Measure the score obtained with the Edinburgh Cognitive and Behavioural Assessment Screen (ECAS) | 24 months
  ECAS is a multidomain assessment questionnaire used in ALS to assess cognitive and behavioural changes where a higher score relates to a better outcome.
Measure the responses in the EQ-5D-5L quality of life health questionnaire. | 24 months
  The EQ-5D-5L questionnaire is a standardised measure of health-related Quality of Life, also incorporating a Visual Analogue Scale. A higher score relates to a better outcome.
Measurement of several biomarkers from blood and urine samples | 24 months
  Urinary P75ECD, plasma neurofilament light and heavy chain, HERV-K expression and genotyping (UNC13a / C9orf72) will be measured for post-trial exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Gold, MD, FFPHM, Principal Investigator — Macquarie University
Locations (28):
- Australia (8):
  - MQ Health Neurology, North Ryde, New South Wales
  - Neuroscience Research Australia (NeuRA), Randwick, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Calvary Health Care Bethlehem, Caulfield South, Victoria
  - The Perron Institute, Nedlands, Western Australia
- Beaumont Hospital, Dublin, Ireland
- UMC Utrecht, Utrecht, Netherlands
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Clinical Trials Unit, Tauranga Hospital, Tauranga
  - Wellington Regional Hospital, Wellington
- Univerzitetni klinični center Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Hospital del Mar, Barcelona
  - Hospital Universitario y Politecnico la Fe, Valencia
- Studiecenheten at Akademiskt specialistcentrum, Stockholm, Sweden
- United Kingdom (10):
  - University of Edinburgh, Anne Rowling Regenerative Nuerology Clinic, Edinburgh
  - The Walton Centre, Liverpool
  - University College London Hospital, London
  - King's College Hospital, London
  - St George's Hospital, London
  - Oxford University Hospital, Oxford
  - Plymouth University Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Sheffield Teaching Hospital, Sheffield
  - Royal Stoke Hotel, Stoke

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated participant level data will be available as open access.
Supporting Information: Study Protocol
Time Frame: Contact the Chief Investigators for access information.
Access Criteria: Contact the Chief Investigators for access information.

REFERENCES:
- [Background] Gold J, Rowe DB, Kiernan MC, Vucic S, Mathers S, van Eijk RPA, Nath A, Garcia Montojo M, Norato G, Santamaria UA, Rogers ML, Malaspina A, Lombardi V, Mehta PR, Westeneng HJ, van den Berg LH, Al-Chalabi A. Safety and tolerability of Triumeq in amyotrophic lateral sclerosis: the Lighthouse trial. Amyotroph Lateral Scler Frontotemporal Degener. 2019 Nov;20(7-8):595-604. doi: 10.1080/21678421.2019.1632899. Epub 2019 Jul 8. PMID 31284774